CLINICAL TRIAL: NCT07301203
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of Single and Multiple Doses of CPD704 Inhalation Suspension in Healthy Chinese Adult Subjects.
Brief Title: Phase I Study of CPD704 Inhalation Suspension in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CPX201-I-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Healthy Participants
Keywords: Phase I Study of CPD704 in Healthy Subjects; CPX201-I-01

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SAD 0.5mg (Other): For SAD 0.5mg cohort will enroll 2 subjects who will receive CPD704 once. 0.5 mg per administration
  Interventions: Drug: CPD704 Inhalation Suspension
- SAD 1.5mg (Other): The SAD 1.5mg cohort plans to enroll 10 subjects with 8 subjects receiving CPD704 and 2 subjects receiving placebo, administered as a single dose per participant.1.5 mg per administration.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- SAD 3mg (Other): This group will include exploratory studies onmetabolite identification, excretion pathways, and excretion quantification(conducted in Cycle 1) as well as anactivated charcoal gastrointestinal absorption blockade study(conducted in Cycle 2). A total of12 subjects will be enrolled (10:2 =CPD704 treatment group: placebo group), Each subject will receive a single 3 mg dose per cycle via oral inhalation.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- SAD 6mg (Other): The SAD 6mg cohort plans to enroll 10 subjects with 8 subjects receiving CPD704 and 2 subjects receiving placebo, administered as a single dose per participant,6 mg per administration.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- SAD 9mg (Other): The SAD 9mg cohort plans to enroll 10 subjects with 8 subjects receiving CPD704 and 2 subjects receiving placebo, administered as a single dose per participant,9 mg per administration.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- SAD 12mg (Other): The SAD 12mg cohort plans to enroll 10 subjects with 8 subjects receiving CPD704 and 2 subjects receiving placebo, administered as a single dose per participant,12 mg per administration..
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- MAD 1.5mg (Other): Each cohort is planned to enroll 12 subjects (10:2 = CPD704 treatment group : placebo group). The route of administration is oral inhalation.
  Based on SAD study results, the MAD cohort will receive QD or BID dosing, with a proposed 5-day consecutive dosing regimen (for BID dosing, only a morning dose will be administered on Day 5, totaling 9 doses).1.5 mg per administration.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- MAD 3mg (Other): Each cohort is planned to enroll 12 subjects (10:2 = CPD704 treatment group : placebo group). The route of administration is oral inhalation.
  Based on SAD study results, the MAD cohort will receive QD or BID dosing, with a proposed 5-day consecutive dosing regimen (for BID dosing, only a morning dose will be administered on Day 5, totaling 9 doses) . 3 mg per administration.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo
- MAD 6mg (Other): Each cohort is planned to enroll 12 subjects (10:2 = CPD704 treatment group : placebo group). The route of administration is oral inhalation.
  Based on SAD study results, the MAD cohort will receive QD or BID dosing, with a proposed 5-day consecutive dosing regimen (for BID dosing, only a morning dose will be administered on Day 5, totaling 9 doses). Each dose:6mg.
  Interventions: Drug: CPD704 Inhalation Suspension; Other: CPD704 placebo

INTERVENTIONS:
Drug: CPD704 Inhalation Suspension — This trial employs standard jet nebulizers (air-compression nebulizers) for oral inhalation administration。
Other: CPD704 placebo — The placebo is administered via standard jet nebulizer (air-compression nebulizer) for oral inhalation
  Arms: MAD 1.5mg; MAD 3mg; MAD 6mg; SAD 1.5mg; SAD 12mg; SAD 3mg; SAD 6mg; SAD 9mg

SUMMARY:
This is a Phase I clinical trial evaluating the safety, tolerability, and pharmacokinetic characteristics of single and multiple doses of CPD704 inhalation suspension in healthy Chinese adult subjects.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled Phase I clinical trial evaluating the safety, tolerability, and pharmacokinetic characteristics of single and multiple doses of CPD704 inhalation suspension administered via nebulization in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject can communicate well with the researchers, fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent form;
2. Healthy subjects aged 18-55 years (including the boundary value, subject to the time of signing the informed consent form), male or female;
3. Body mass index (BMI) within the range of 19 ~ 28 kg/m2 (including the critical value), male weight ≥ 50 kg, female weight ≥ 45 kg;
4. The subject has no plans to give birth, sperm or egg donation from the signing of the informed consent form to 90 days after medication, and voluntarily takes medically approved contraceptive measures (including his partner)

Exclusion Criteria:

1. Patients who have taken any clinical trial drugs or participated in any drug clinical trial within 3 months before signing the ICF, or participated in other medical research activities, and are not suitable for participating in this trial as judged by the investigator;
2. Previous or combined with the following diseases, cardiovascular disease [such as heart failure (such as fluid retention and edema), unstable ischemic heart disease, congestive heart failure poor control of coronary artery disease, myocardial infarction, long QT syndrome history, etc.], respiratory, renal, neurological, endocrine, immune, skin, gastrointestinal (such as gastrointestinal ulcers or gastrointestinal bleeding, etc.), liver or blood system and other diseases/abnormal history, the investigators judge that their participation in this trial may affect the safety of subjects or affect the analysis of study results;
3. Patients with the following mental illness: 1) Uncontrolled/unstable major depressive disorder (MDD) or other serious mental disorders (such as schizophrenia, bipolar disorder or other serious mood or anxiety disorders) within 2 years before screening; 2) Suicide attempt or suicidal behavior 30 times before screening; 3) Suicidal ideation corresponding to Columbia-Suicide Severity Rating Scale (C-SSRS) category 4 or 5 in the past 30;
4. Known hypersensitivity, immune reaction or intolerance to CPD704 Inhalation Suspension or any of the excipients in the drug product (polysorbate 80, sodium chloride, sodium citrate dihydrate, disodium edetate, sodium hydroxide or hydrochloric acid) and/or unsuitable for treatment with CPD704 Inhalation Suspension;
5. Long-term oral drugs can not be stopped or suffering from gastric ulcer, gastritis affecting oral activated charcoal, or allergic to activated charcoal;
6. Patients with severe infection, trauma or major surgery before signing the ICF, or planning to undergo surgery during the trial;
7. Use of any live vaccines (except influenza vaccine) within 28 days before signing the ICF or plan to receive vaccines during the study;
8. Blood loss or blood donation of more than 400 mL within 3 months before signing the ICF (excluding female menstrual blood loss), or intend to donate blood during the trial or within 1 month after the end of the trial;
9. Smokers or those who smoke more than 5 cigarettes per day within 3 months before signing the ICF, or those who cannot comply with the provisions of prohibiting smoking during the trial, or those who test positive for urine cotinine;
10. Pulmonary ventilation function test Forced expiratory volume in the first second (FEV1) measured value/FEV1 predicted value ≤ 80% or forced vital capacity (FVC) ≤ 80% of predicted value or any other clinically significant abnormalities;
11. Use of any drugs that inhibit or induce hepatic drug-metabolizing enzymes within 28 days before signing the ICF; or use of any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products within 14 days before signing the ICF. If the half-life of concomitant drugs is increased, the required time interval should be at least 5 half-lives of the drug;
12. Excessive consumption of tea, coffee or caffeinated beverages (an average of more than 8 cups per day, 250 mL per cup) within 6 months before signing the ICF;
13. Consumption of any grapefruit, caffeine-containing beverages or foods (such as grapefruit juice, coffee, strong tea, chocolate, caffeine-containing carbonated beverages, cola, cocoa, etc.) within 48 hours before the first dose;
14. Those who have special requirements for diet and cannot abide by the unified diet;
15. Unwilling or unable to tolerate multiple venipuncture or difficult venous blood sampling or a history of fainting;
16. Previous history of drug abuse/drug use, or drug abuse screening (including tetrahydrocannabinolic acid, morphine, ketamine, methamphetamine, benzodiazepine, cocaine) results were positive;
17. Regular drinking within 6 months before signing the ICF [i.e., women drink more than 14 standard units of alcohol per week, men drink more than 21 standard units of alcohol per week (1 standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine)] or can not abstain from alcohol during the trial; or positive breath alcohol test;
18. The results of physical examination, vital signs examination, ECG, laboratory tests (blood routine, blood biochemistry, coagulation function, thyroid function, urine routine, stool routine, etc.), chest X-ray, abdominal B ultrasound examination during the screening period are judged by the study doctor as abnormal and clinically significant;
19. Abnormal ECG findings during the screening period, such as bradycardia or tachycardia (heart rate < 50 bpm or > 100 bpm), QTc prolongation (QTcF interval ≥ 450 ms in males and ≥ 470 ms in females, corrected according to Fridericia's formula), arrhythmia, etc., and clinically significant as judged by the investigator;
20. Patients with positive results of any test of hepatitis B surface antigen (HbsAg), hepatitis C virus antibody (HCV-Ab), treponema pallidum antibody (Syphilis TP) and human immunodeficiency virus test (HIV-Ag/Ab) during the screening period;
21. Pregnant or lactating women, or positive blood pregnancy test results;
22. Unwilling or unable to correctly use the nebulizer according to the nebulizer instructions Inhalation of investigational drugs or nebulizer use training failed;
23. Any other condition that, in the opinion of the investigator, would make participation in the study inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-07-18 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes | From the date of informed consent signature until Day 7 for SAD group(Day 14 for SAD 3mg group) and Day 11 for MAD Group.
  Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after first dose
  Plasma concentrations of CPD704 following nebulization of CPD704 inhalation suspension
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after last dose
  Cmax of CPD704 following nebulized administration of CPD704 inhalation suspension
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after last dose
  Time to reach peak plasma concentration (Tmax) of CPD704 following nebulized administration of CPD704 inhalation suspension
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after last dose
  Area under the plasma concentration-time curve from time zero to time t (AUC0-t) of CPD704 following nebulized administration of CPD704 inhalation suspension
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after last dose
  t1/2 of CPD704 after nebulization of CPD704 inhalation suspension
Pharmacokinetic (PK) endpoints | During the period starting 60 minutes before initial drug administration through to 48hours after last dose
  PK profile of CPD704 inhalation suspension following activated charcoal blockade (including AUC0-∞, AUC0-t, Cmax and other parameters)

OTHER OUTCOMES:
QTcF interval | From 60 minutes prior to first dose until 12 hours of first dose.
  Evaluation of QTcF interval prolongation potential following single-dose administration of CPD704 inhalation suspension in healthy adult volunteers
Metabolites and excretion pathways | only applicable for SAD 3mg cohort, From 60 minutes prior to first dose until 48Hours of last dose.
  Preliminary investigation of CPD704 metabolites in humans and primary excretion pathways, including cumulative excretion rates of the parent drug and metabolites (if applicable) in urine and feces

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided